CLINICAL TRIAL: NCT05293184
Title: The Global Angelman Syndrome Registry
Acronym: GASR
Status: Recruiting | Type: Observational
Sponsor: Foundation for Angelman Syndrome Therapeutics, Australia (Other)
Collaborators: Queensland University of Technology (Other)
Responsible Party: Principal Investigator, Associate Professor Helen (Honey) Heussler, Associate Professor, Paediatrics and Child Health, The University of Queensland
Other Study IDs: RG-16-078-AM01
Record Dates: First submitted 2017-06-27; First posted 2022-03-24 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Angelman Syndrome
Keywords: Angelman Syndrome; Registries; Observational study only
MeSH Terms: conditions — Angelman Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 70 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with Angelman Syndrome: Individuals from birth to adulthood with Angelman Syndrome
  Interventions: Other: Observational study only

INTERVENTIONS:
Other: Observational study only

SUMMARY:
The Global Angelman Syndrome Registry is an online patient organisation driven registry to collect information about the natural history of children and adults with Angelman Syndrome. The registry will facilitate 1) recruitment for clinical trials into therapies and interventions to benefit participants with Angelman Syndrome and their families, and 2) advancement of research and best standards of care for Angelman Syndrome.

The registry is currently available in English, Spanish, Traditional Chinese, Italian, Polish, Hindi, and Brazilian Portuguese.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Angelman Syndrome

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a diagnosis of Angelman Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-09-28 (Actual); Primary Completion 2099-12-31 (Estimated); Study Completion 2099-12-31 (Estimated)

PRIMARY OUTCOMES:
Gather longitudinal data on individuals living with Angelman Syndrome | 70 years (lifespan)
  Parent/ caregiver reporting on diagnosis, clinical status, and patient-reported outcomes of individual living with Angelman Syndrome. This will be achieved by inviting parents/ caregivers with additional questionnaire like modules, and tracking changes in their responses over time.

CONTACTS AND LOCATIONS:
Overall Officials: Helen (Honey) Heussler, MBBS, FRACP DM, Principal Investigator — The University of Queensland
Locations (1):
- Queensland University of Technology, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Yes
All external researchers wishing to recruit registry participants for clinical trials or access data are encouraged to review the information on our website (https://www.angelmanregistry.info/collaborate-with-us/) and contact the data curator (curator@angelmanregistry.info)
Supporting Information: Study Protocol, ICF
Time Frame: Duration of project.
Access Criteria: External researchers wishing to access registry data or recruit participants must comply with the directions outlined above.
URL: https://angelmanregistry.info

REFERENCES:
- [Background] Napier KR, Tones M, Simons C, Heussler H, Hunter AA, Cross M, Bellgard MI. A web-based, patient driven registry for Angelman syndrome: the global Angelman syndrome registry. Orphanet J Rare Dis. 2017 Aug 1;12(1):134. doi: 10.1186/s13023-017-0686-1. PMID 28764722
- [Background] Tones M, Cross M, Simons C, Napier KR, Hunter A, Bellgard MI, Heussler H. Research protocol: The initiation, design and establishment of the Global Angelman Syndrome Registry. J Intellect Disabil Res. 2018 May;62(5):431-443. doi: 10.1111/jir.12482. PMID 29633452
- [Background] Tones M, Zeps N, Wyborn Y, Smith A, Barrero RA, Heussler H, Cross M, McGree J, Bellgard M. Does the registry speak your language? A case study of the Global Angelman Syndrome Registry. Orphanet J Rare Dis. 2023 Oct 19;18(1):330. doi: 10.1186/s13023-023-02904-1. PMID 37858180
- [Result] Roche, L., Tones, M., Williams, M.G. et al. Caregivers Report on the Pathway to a Formal Diagnosis of Angelman Syndrome: A Comparison Across Genetic Etiologies within the Global Angelman Syndrome Registry. Adv Neurodev Disord 5, 193-203 (2021). https://doi.org/10.1007/s41252-021-00195-w
- [Result] Leader G, Whelan S, Chonaill NN, Coyne R, Tones M, Heussler H, Bellgard M, Mannion A. Association between early and current gastro-intestinal symptoms and co-morbidities in children and adolescents with Angelman syndrome. J Intellect Disabil Res. 2022 Nov;66(11):865-879. doi: 10.1111/jir.12975. Epub 2022 Sep 2. PMID 36052644
- [Result] Roche, L., Tones, M., Cross, M. et al. An Overview of the Adaptive Behaviour Profile in Young Children with Angelman Syndrome: Insights from the Global Angelman Syndrome Registry. Adv Neurodev Disord 6, 442-455 (2022). https://doi.org/10.1007/s41252-022-00278-2
- [Result] Leader G, Gilligan R, Whelan S, Coyne R, Caher A, White K, Traina I, Muchenje S, Machaka RL, Mannion A. Relationships between challenging behavior and gastrointestinal symptoms, sleep problems, and internalizing and externalizing symptoms in children and adolescents with Angelman syndrome. Res Dev Disabil. 2022 Sep;128:104293. doi: 10.1016/j.ridd.2022.104293. Epub 2022 Jul 4. PMID 35797778

DOCUMENTS (1):
  • Informed Consent Form (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT05293184/ICF_000.pdf